CLINICAL TRIAL: NCT02334111
Title: Project RESPECT-Plus: Recovery, Empowerment, Social Services, Prenatal Care, Education and Community Treatment-Plus
Brief Title: RESPECT-PLUS: Services for Infants With Prenatal Opiate Exposure
Acronym: RESPECT-Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Ruth Rose-Jacobs Sc.D., Associate Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HHS-2012-ACF-ACYF-CB-0286
Record Dates: First submitted 2014-04-15; First posted 2015-01-08 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Opioid Use Disorder; Neonatal Abstinence Syndrome; Child Development; Child Abuse; Child Neglect
Keywords: Parenting Support for Mothers in Recovery; Neonatal Abstinence Syndrome; Social Determinants of Health; Child Development; Child Abuse; Child Neglect; Primary Care
MeSH Terms: conditions — Opioid-Related Disorders; Neonatal Abstinence Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- (Control) (No Intervention): Patients will receive standard of care
- (Intervention) (Experimental): Patients will receive RESPECT-Plus intervention
  Interventions: Behavioral: RESPECT-Plus

INTERVENTIONS:
Behavioral: RESPECT-Plus — A RESPECT-Plus family specialist (FS) will deliver the intervention to subjects (mothers in treatment for opiate use disorder) recruited during their third trimester of pregnancy and randomized into the study's intervention arm post-delivery. During their infant's hospital stay, the FS will schedule a convenient time to meet the subjects (mothers) to educate them on infant soothing techniques. With permission from the mother, the FS will join the subjects during their infant's routine well-child visits at the pediatric primary site. Optional home visiting provides another meeting opportunity between the subjects and FS.
  Arms: (Intervention)

SUMMARY:
The impact of parental opioid use disorder and other substance use exposure on child welfare and the healthcare system is undeniable. Between 2000 and 2009, the number of delivering mothers using or dependent on opiates rose nearly five-fold, and it is estimated that 48-94% of children exposed to opioids in utero will be diagnosed with neonatal abstinence syndrome (NAS), a set of behavioral and physiological complications resulting from abrupt substance withdrawal at birth. Opioid abuse is usually coupled with use of other substances, and research has demonstrated that children born to parents with substance use disorders are three to four times more likely to suffer abuse or neglect.

Currently, the standard of care for pregnant women who are being treated for opiate dependence at Boston Medical Center (BMC) is to receive all their prenatal care in the RESPECT Clinic, an innovative program of the BMC Department of Obstetrics and Gynecology designed to treat addiction during the prenatal and early postnatal period. Once the child is born, BMC staff files a report of suspected child abuse and neglect in accordance with the Massachusetts General Laws section 51A. The state Department of Children and Families makes a determination regarding the disposition of these families. Medically, most of these children are treated in-patient at BMC for NAS and then discharged to follow-up with routine pediatric primary care. Currently, approximately 85% of infants born exposed to opioids go home with their mothers, and the remainder receive substitute care, either with other family members or via foster care.

This investigation is a randomized controlled trial of RESPECT-Plus, a continuum of promising and evidence-based practices designed to strengthen family protective factors and improve health permanency and well-being outcomes for children born to mothers in treatment for opioid use disorder. Anticipated outcomes of the intervention include fewer reports of supported child abuse or neglect filings in the child's first year of life, fewer days in out-of-home placement; fewer terminations of parental rights in the child's first year of life; and improvements in family functions overall (e.g. improved access to basic needs/social determinants of health, improved parental resilience, and decreased maternal depression).

DETAILED DESCRIPTION:
Project RESPECT-Plus (Recovery, Empowerment, Social Services, Prenatal care, Education, and Community Treatment-Plus) is a randomized controlled trial of promising and evidence-based practices designed to strengthen family protective factors and improve health permanency and well-being outcomes for children born to mothers in treatment for opioid use disorder. The target population for project RESPECT-Plus is pregnant women in treatment for opiate use disorder receiving prenatal care at BMC's RESPECT Clinic. A total of 200 subjects - 100 mothers - will be enrolled into the study and randomized post-partum to receive the intervention or standard of care, and will be followed for 1 year.

In order to provide continuity of care from the prenatal to pediatric primary care setting, participants receiving prenatal care at the RESPECT Clinic are recruited during their third trimester of pregnancy. After consent, the initial baseline data collection is scheduled and once the infants are born and pass the eligibility screening (term birth and no major congenital abnormalities or developmental disabilities), mothers and their infants are randomized into the intervention (RESPECT-Plus) or control (standard of care) group.

The intervention is delivered by a family specialist who, with the permission of the mother, will attend routine well-child visits so as to collaborate with providers in the child's medical home and parent through the medical visit. As desired by the mother, home visits, other face-to-face contacts, telephone calls, and text messages will assist in addressing social determinants of health, improve the mother's knowledge of child development and parenting, and link families to community resources to address existing concrete support needs. The family specialist will receive support and training by a licensed clinical social worker and the Medical-Legal Partnership, Boston (MLP Boston) to identify legal and social needs that may affect a child's health and development and to take action either by helping family members advocate for themselves, or by referring them to an appropriate public health, legal, or social service agency or resources.

Both the intervention and standard of care groups will be evaluated by research evaluators not associated with the intervention at baseline, and when the child is 6 and 12 months old.

The two goals and associated objectives for RESPECT-Plus are:

1. To evaluate the RESPECT-Plus intervention, on improving child well-being, safety, and permanency outcomes.
2. To evaluate family functioning aligned with the five protective factors in the Strengthening Families model (parental resilience, knowledge of parenting and child development, concrete supports, social connections, and child factors).

Anticipated outcomes of the intervention include fewer reports of supported child abuse or neglect filings in the child's first year of life, fewer days in out-of-home placement and terminations of parental rights in the child's first year of life, and improvements in family functions overall (e.g. improved access to basic needs/social determinants of health, improved parental resilience, and decreased maternal depression).

ELIGIBILITY:
Inclusion Criteria:

1. Opiate-dependent pregnant women receiving opiate-replacement therapy (methadone or buprenorphine) treatment by licensed provider (mother)
2. Receives prenatal and obstetric care through Boston Medical Center's RESPECT clinic (mother)
3. Due date within 3 months at time of enrollment (Estimated Gestation Age >27 weeks) (mother)
4. 18 years and older (mother)
5. Singleton pregnancy (infant)
6. Intends to deliver at Boston Medical Center (mother)
7. Intends to remain in the Boston area after birth of child (mother)
8. Mother able to provide informed consent (not excluded by RESPECT staff)
9. No serious medical illness in infant such as sepsis, asphyxia, seizures, or respiratory failure (infant)
10. No major congenital abnormalities in infant including genetic syndromes (infant)
11. Gestational age at birth 36 weeks or greater defined by obstetrical estimate (infant)
12. Born at Boston Medical Center (infant)
13. Not incarcerated at the time of enrollment (mother)

Exclusion Criteria:

1. Plans to voluntarily relinquish parental rights at birth
2. Does not speak English.
3. Estimated gestational age less than 36 weeks
4. Infant positive for serious congenital anomaly or developmental disability

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to Change in Custody | up to 12 months post-birth
  Child welfare data will be obtained for all enrolled infant subjects from the Department of Children and Families (DCF). DCF will provide information concerning any changes in custody. The study outcome will be time to change in custody as primary outcome.

SECONDARY OUTCOMES:
Improvements in parental resilience and parenting aligned with the Strengthening Families model (parental resilience, knowledge of parenting and child development, concrete supports, social connections, and child well-being) | Outcomes will be measured at baseline, 6 months, and 12 months (child-related measures only administered at 6 and 12 months post-birth)
  This composite measure involves evaluating important factors associated with parenting. This will include the Edinburgh Post-natal Depression Scale, the Connor-Davidson Resilience Scale, the Difficult Life Circumstances Scale, the Inventory of Socially Supportive Behaviors, and additional measures to assess material hardships and access to public assistance programs.

OTHER OUTCOMES:
Process Data | Measures will be taken at 6 and 12 months
  This composite measure involves examining patient-reported information on services received, such as SNAP (Special Supplemental Nutrition Program for Women, Infants, and Children), etc and documentation from Family Specialists on support services given during the Family Specialist encounters including phone, in person, coordinated primary care visits, and home visits (if applicable). The time devoted to the care of each participating family will be collected and collated. This data collection will be documented in a Microsoft Access database.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Rose-Jacobs, Sc.D., Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No